CLINICAL TRIAL: NCT04262011
Title: Effect of Non-surgical Periodontal Treatment on Renal Function and C-reactive Protein Levels in Hemodialysis Patients
Brief Title: Effect of Non-surgical Periodontal Treatment and C-reactive Protein Levels in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Fabricio Batistin Zanatta, Principal advisor, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10453519.4.0000.5346
Record Dates: First submitted 2019-12-17; First posted 2020-02-10 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Chronic Kidney Disease Stage 5; Periodontitis
Keywords: chronic kidney disease; hemodialysis; periodontal diseases; periodontitis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Periodontitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: The study will have two groups, one receiving immediate periodontal treatment and the other receiving late periodontal treatment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to the group to which the patient belongs, whether immediate or late.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate treatment (Other): After randomization, patients who are allocated to the immediate treatment group will receive treatment.
  Interventions: Procedure: immediate treatment
- postponed treatment (Other): After randomized patients will be allocated to this group, they will wait for the follow-up of the study to receive delayed treatment.
  Interventions: Procedure: postponed treatment

INTERVENTIONS:
Procedure: immediate treatment — Patients allocated to the immediate treatment group will receive full mouth treatment, and will use 0.12% chlorhexidine mouthwash, every 12 hours for a week, and will receive oral hygiene instructions throughout the follow-up period. Patients will be evaluated at the beginning, at 3 and 6 months.
  Arms: immediate treatment
Procedure: postponed treatment — Patients allocated to the late treatment group will be assessed at baseline, 3 and 6 months. After the end of the follow-up period, they will receive non-surgical periodontal treatment performed in four sessions.
  Arms: postponed treatment

SUMMARY:
The presence of periodontitis has been hypothesized as a risk factor for several systemic outcomes, including chronic kidney disease (CKD). Therefore, the aim of this study is to evaluate the impact of non-surgical periodontal treatment on CRP levels and quality of life of patients with chronic kidney disease undergoing hemodialysis (HD) in Santa Maria-RS.

DETAILED DESCRIPTION:
C-reactive protein (CRP) has been identified as a possible mediator of the association between periodontitis and various systemic diseases. The presence of periodontitis has been hypothesized as a risk factor for several systemic outcomes, including chronic kidney disease (CKD). Therefore, the aim of this study is to evaluate the impact of non-surgical periodontal treatment on CRP levels and quality of life of patients with chronic kidney disease undergoing hemodialysis (HD) in Santa Maria-RS. A total of 88 patients with severe periodontitis who are on HD therapy will be included in this study. At baseline, periodontal, radiographic, blood test, and quality-of-life questionnaire will be assessed for all patients, after which severe periodontitis will be defined according to the American Association of Periodontology and European Federation of Periodontology. The 88 patients with periodontal disease will be randomized and divided into two groups. One group will receive full mouth non-surgical periodontal treatment (TPNC) and a late treatment group that will receive TPNC only at the end of the study. All patients will receive follow-up of periodontal parameters and blood collection for initial CRP assessment at 3 and 6 months after treatment. Outcome evaluators will be blind to the group the patient belongs to. Patients in the immediate treatment group will receive follow-up oral hygiene instructions and use 0.12% chlorhexidine mouthwash during the first week after treatment.

ELIGIBILITY:
Minimum Age: 18 Years Sex: All Accepts Healthy Volunteers: No

Criteria:

Inclusion Criteria:

* Having been diagnosed with chronic kidney disease (CKD) for at least 90 days.
* Have at least 8 teeth in the mouth.
* For the patient to be classified as having periodontal disease, he must have at least two nonadjacent sites with insertion loss of 3mm or more and two nonadjacent sites with probing depth of 4mm or more.

Exclusion Criteria:

Ineligible individuals were characterized by exhibiting one of the following conditions:

* Patients diagnosed with malignant neoplasia;
* Patients diagnosed with carriers of the HIV virus;
* Pregnant or lactating women;
* Patients with absence of all dental elements (total edentulous);
* Patients undergoing orthodontic treatment;
* Patients who have received periodontal treatment in the last 6 months.
* Patients with active infection (other than periodontitis) who require antibiotic prophylaxis;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-02-29 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
effect of periodontal treatment on levels of systemic inflammatory markers | baseline changes by 6 months follow-up
  To evaluate the impacts of periodontal treatment on the levels of systemic inflammatory markers such as C-reactive protein, albumin and transferrin saturation. The patients will be submitted to the collection of blood sample in the baseline, 3 and 6 months to obtain the clinical variables.

SECONDARY OUTCOMES:
effect of periodontal treatment on oral health-related quality of life | baseline changes by 6 months follow-up
  To assess the impacts of periodontal treatment on overall quality of life and oral health that will be assessed using the questionnaire Oral Health Impact Profile (OHIP14) (14 items), in this questionnaire the higher the score, the worse the quality of life is considered.
effect of periodontal treatment on overall quality of life | baseline changes by 6 months follow-up
  To assess the impacts of periodontal treatment on overall quality of life and oral health that will be assessed using the questionnaire The Short-Form Health Survey (SF-36) (36 items). In this questionnaires, the higher the score, the worse the quality of life is considered.
effect of periodontal treatment on overall quality of life and related to kidney disease | baseline changes by 6 months follow-up
  o assess the impacts of periodontal treatment on overall quality of life and oral health that will be assessed using the questionnaire Kidney Disease Quality of Life Short Form (KDQOL-SF) (80 items). This scale ranges from 0 to 100, higher values show a better quality of life.
effect of periodontal treatment on psychological condition in patients with chronic kidney disease undergoing hemodialysis | baseline changes by 6 months follow-up
  ndividuals' psychological condition will be assessed using the Depression - Anxiety - Stress Scale 21 (DASS 21) (21 items).The highest grades in each scale correspond to more negative affective states.
effect of periodontal treatment on psychological condition | baseline changes by 6 months follow-up
  Individuals' psychological condition will be assessed using the sense of coherence (SOC 13) which proposes to explain successful strategies to cope with stress. For the final score calculation, the items are summed and the result can vary from 13 to 65, where higher scores represent SOC. The the greater the result, the greater the coping capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel P Antoniazzi, pHD, Study Director — Universidade Federal de Santa Maria; Samantha S Santi, DS, Study Chair — Universidade Federal de Santa Maria; Leandro M Oliveira, MS, Study Chair — Universidade Federal de Santa Maria; Rafaela V Palmeira, MS, Study Chair — Universidade Federal de Santa Maria; Catiusse C Del'Agnese, MS, Study Chair — Universidade Federal de Santa Maria
Locations (1):
- Fabricio Batistin Zanatta, Santa Maria, Rua Floriano Peixoto--, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang F, Wu B, Qu Q, Gao J, Yan W, Huang X, Ma D, Yue J, Chen T, Liu F, Liu Y. The clinical response and systemic effects of non-surgical periodontal therapy in end-stage renal disease patients: a 6-month randomized controlled clinical trial. J Clin Periodontol. 2015 Jun;42(6):537-46. doi: 10.1111/jcpe.12411. Epub 2015 May 30. PMID 25933364